CLINICAL TRIAL: NCT07265752
Title: Tirzepatide for the Treatment of Cannabis Use Disorder: A Pilot Double-blind, Placebo-controlled, Crossover Trial
Brief Title: Tirzepatide for the Treatment of Cannabis Use Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joji Suzuki, MD, Principal Investigator, Division of Addiction Treatment and Prevention, AMC Psychiatry Mass General Brigham, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P002984
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cannabis Use Disorder
Keywords: tirzepatide
MeSH Terms: interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- tirzepatide (Experimental): 2.5mg subcutaneous injection once
  Interventions: Drug: Tirzepatide
- placebo (Placebo Comparator): matching placebo subcutaneous injection once
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — 2.5mg subcutaneous injection once
  Arms: tirzepatide
Drug: Placebo — Saline placebo subcutaneous injection once
  Arms: placebo

SUMMARY:
This is a pilot randomized cross-over trial to examine the effects of tirzepatide on cue-reactivity among individuals with cannabis use disorder.

DETAILED DESCRIPTION:
This is a pilot randomized cross-over trial to examine the effects of tirzepatide on cue-reactivity among individuals with cannabis use disorder. Eligible participants will be scheduled in random order to receive either tirzepatide or placebo injection in double-blind fashion and cross-over design. Outcomes will be assessed at the following study visit. Washout period of at least 4 weeks will be required between tirzepatide or placebo injections. Primary outcome of interest is cue-induced craving to cannabis-related visual cues.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults aged 18 and above
* Diagnosed with DSM-5 cannabis use disorder, severe

Exclusion Criteria:

* Active psychosis, active suicidality or homicidality or any psychiatric condition that impair ability to provide informed consent
* Any current or lifetime diagnosis of eating disorders including anorexia, bulimia, binge eating or
* Comorbid substance use disorder
* BMI<21 kg/m2
* Current or lifetime diagnosis of Type 1 or Type 2 diabetes
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
* Use of any glucagon-like peptide -1 agonist medications in the prior 3 months
* Anticipating receipt of any glucagon-like peptide-1 agonist medications during the trial
* Current hypoglycemia as indicated by a blood sugar level of <71 mg/dL measured at baseline visit, as well as visits 2 and 4.
* Untreated cholelithiasis or gallbladder disease
* History of acute myocardial infarction, cerebrovascular accident (stroke), unstable angina, or congestive heart failure in the last 90 days
* Systolic blood pressure persistently above 160 mmHg or diastolic blood pressure persistently above 100 mmHg during screening
* History of inflammatory bowel disease, bariatric surgery, pancreatitis, diabetic gastroparesis, or non-arteritic anterior ischemic optic neuropathy
* Liver function test greater than 3 times upper normal limit
* Renal impairment as indicated by estimated glomerular filtration rate (eGFR) of <30
* History of hypersensitivity or allergy to tirzepatide
* Pregnant or breastfeeding
* Individuals taking glucagon-like peptide-1 agonists or other weight loss drugs.
* Anticipated to participate in a concurrent drug trial
* Any other reason or clinical condition that the investigators judge may interfere with study participation and/or be unsafe for a participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Cue-Induced Craving | 5 weeks
  Craving scores will be assessed using a cue-reactivity paradigm in which participants are exposed to cannabis]-related cues. Scores range from 0 to 30, with higher scores indicating greater craving intensity.

SECONDARY OUTCOMES:
Serious adverse event | 5 weeks
  Incidence of serious adverse events
Cravings | 5 weeks
  Cannabis craving scale using the 12-item questionnaire, each item scored on a 1-7 sale. Higher scores (either average or summed) indicates stronger cravings.
Abstinence | 5 weeks
  Percent days abstinent from cannabis
Weight | 5 weeks
  Weight
Blood sugar | 5 weeks
  Blood glucose
Hemoglobin A1c | 5 weeks
  Hemoglobin A1c
Depression severity as measured by the Patient Health Questionnaire-8 (PHQ-8) | 5 weeks
  Depression severity as measured by the Patient Health Questionnaire-8 (PHQ-8). The PHQ-8 assesses depression severity over the past two weeks. Total scores range from 0 to 24, with higher scores indicating greater depression severity (worse outcome). Score interpretation: 0-4 (none), 5-9 (mild), 10-14 (moderate), 15-19 (moderately severe), 20-24 (severe depression).
Anxiety severity as measured by the Generalized Anxiety Disorder-7 scale (GAD-7) | 5 weeks
  The GAD-7 assesses anxiety symptom severity over the past two weeks. Total scores range from 0 to 21, with higher scores indicating greater anxiety severity (worse outcome). Score interpretation: 0-4 (minimal anxiety), 5-9 (mild), 10-14 (moderate), 15-21 (severe anxiety).
Suicidality as measured by the C-SSRS (Columbia-Suicide Severity Rating Scale) | 5 weeks
  The C-SSRS assesses the presence and severity of suicidal ideation and behavior. Suicidal ideation severity scores range from 0 to 5 (0=no ideation, 1=wish to be dead, 2=non-specific active suicidal thoughts, 3=active suicidal ideation with methods, 4=suicidal intent, 5=suicidal intent with plan), with higher scores indicating greater severity (worse outcome). The scale also captures suicidal behavior as binary yes/no responses.

CONTACTS AND LOCATIONS:
Overall Officials: Joji Suzuki, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No